CLINICAL TRIAL: NCT05258643
Title: The Role of Natural Killer, Complement and T-lymphocytes in COVID-19 Disease, a Prospective Monocentric Study
Acronym: TONIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020/177
Record Dates: First submitted 2021-11-03; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2021-04

CONDITIONS: Complement Abnormality; Peripheral Blood Mononuclear Cells; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Covid-19 patients (Other): Whole blood and serum samples will be collected during acute disease (inclusion and 7 days after inclusion) and during patient follow-up at 2 months after infection
  Interventions: Other: Blood analysis
- Controle (Other): Whole blood and serum samples will be collected during the same period
  Interventions: Other: Blood analysis

INTERVENTIONS:
Other: Blood analysis — Venipuncture and collection of serum and whole blood

SUMMARY:
The current study is an open, non-randomized, monocentric, and interventional study. CoViD-19 patients will be recruited at UZ Brussel after informed consent is obtained. Whole blood and serum samples will be collected during acute disease (inclusion and 7 days after inclusion) and during patient follow-up at 2 months after infection.

Sample storage and subsequent use in fundamental research will be performed at VUB Neuro-Aging and Viro-Immunotherapy.

Additionally, medical records of UZ Brussel will be searched and epidemiological, clinical, radiological, and biological data of the selected patients will be obtained at the diagnosis time point and during follow-up.

Healthy volunteers will be recruited as well in the current study, as a comparison arm, after informed consent is obtained.

ELIGIBILITY:
Covid-19 patients

Inclusion Criteria:

* Positive nasopharyngeal reverse transcriptase-polymerase chain reaction for SARS-Coronavirus-02
* Signed inform consent

Healthy Volunteers

Inclusion Criteria:

* Signed inform consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in complements or peripheral blood mononuclear cells between CoViD-19 patients and controls | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Allard, PhD, Study Director — UZ Brussel (Vrije Universiteit Brussel); Joeri Aerts, PhD, Study Chair — Vrije Universiteit Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided